CLINICAL TRIAL: NCT00478179
Title: A Randomized, Double-Blind, Placebo Controlled, Two-Way Cross-Over Study of Analgesic Efficacy of Bupivacaine Transdermal Therapeutic System in Patients With Post-Herpetic Neuralgia
Brief Title: Study of a Bupivacaine Patch (Eladur™) to Treat Post- Herpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durect (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN005-0009
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Postherpetic Neuralgia; Pain
Keywords: herpes zoster; shingles; PHN; post herpetic neuralgia; neuropathic pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Pain; Herpes Zoster; Neuralgia | interventions — Administration, Cutaneous; Transdermal Patch

INTERVENTIONS:
Drug: Transdermal/Patch (Bupivacaine TTS [Eladur™])

SUMMARY:
Neuropathic pain is caused by a virus commonly associated with chicken pox. This virus may become dormant in the nervous system and later reactivate causing herpes zoster, also known as "shingles". Post-herpetic neuralgia (PHN) is a persistent pain in the area of healed skin lesions. This study will test the safety and efficacy of treating PHN patients with the analgesic patch, Bupivacaine TTS (Eladur™).

ELIGIBILITY:
Inclusion Criteria:

* Male or females age 21 years or older.
* Pain in thoracic or lumbar regions for a minimum of 90 days after crusting of Herpes Zoster (HZ) lesions.
* Stable prescribed medications regimen (including opioids, anticonvulsants, and tricyclic antidepressants).
* Intact, unbroken skin over the painful area to be treated.
* Body Mass Index (BMI) no more than 35 kg/m2.

Exclusion Criteria:

* Active HZ lesions, dermatitis, Central Nervous System (CNS) injury.
* Any immunosuppressed condition, including but not limited to AIDS/HIV and Hodgkin's lymphoma.
* Pain control by nerve block or neurosurgical intervention.
* Evidence of clinically significant hepatic, gastrointestinal, renal, hematologic, urologic, neurologic, respiratory, endocrine or cardiovascular system abnormalities, psychiatric disorders, or acute infection.
* Connective tissue disorders (systemic lupus erythematosus, scleroderma, mixed connective tissue disease).
* Recent use (within 30 days preceding the first treatment visit) of any topically applied pain medication, such as nonsteroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics (including Lidoderm®), steroids or capsaicin products on the painful areas.
* Significant pain of an etiology other than PHN, for example, compression-related neuropathies (e.g., spinal stenosis), fibromyalgia or arthritis. Patients must not have significant ongoing pain from other cause(s) that may interfere with judging PHN related pain.
* Participation in a clinical trial of an investigational product or device within 30 days of the screening visit or concurrently during the conduct of this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Reduction of pain with mean daily pain intensity

SECONDARY OUTCOMES:
Subject's satisfaction of treatment; Change in neuropathic pain; Patch adherence.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - La Jolla, California
  - Loma Linda, California
  - Santa Monica, California
  - Bradenton, Florida
  - Altoona, Pennsylvania
  - Salt Lake City, Utah
  - Tacoma, Washington